CLINICAL TRIAL: NCT00749346
Title: An Open Label Pilot Study of NovoTTF-100L in Combination With Pemetrexed (Alimta®) for Advanced Non-small Cell Lung Cancer
Brief Title: NovoTTF-100L in Combination With Pemetrexed (Alimta®) for Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EF-15
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Non-small Cell Lung Cancer; NSCLC
Keywords: TTFields; NSCLC; Alimta; Pemetrexed
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Treatment with concomitant Alimta and NovoTTF-100L
  Interventions: Device: NovoTTF-100L

INTERVENTIONS:
Device: NovoTTF-100L — TTFields treatment 12h/d for the duration of the study (until progression)concomitant to standard Alimta dosing
  Other Names: TTFields; Pemetrexed; Alimta; Electric fields

SUMMARY:
An open-label phase I-II trial will be performed in 42 patients with pretreated locally advanced non-small cell lung cancer. The trial is designed to estimate the efficacy and to determine safety of NovoTTF-100L treatment combined with Pemetrexed for advanced NSCLC patients. Patients will receive standard Pemetrexed therapy (at 500 mg/m2 iv q3w for 3 cycles) concomitant to NovoTTF-100L therapy (12 hours a day, daily until the end of all three cycles of Alimta). Repeat treatments with Alimta + NovoTTF-100L will be offered as long as the patient is stable or responding. If there is a in-field response with progression outside of the NovoTTF field, Pemetrexed is to be stopped and third line chemotherapy with Docetaxel is to be initiated (35 mg/m2 weekly, d1, 8, 15, q 28 d).

DETAILED DESCRIPTION:
The trial will be conducted in two stages. Fourteen patients will be recruited to a phase I stage of the trial. After all 14 patients have received 3 courses of Alimta (9 weeks of NovoTTF-100L treatment), these patients will be analyzed for toxicity. If the incidence of device related serious adverse events is < 20%, the trial will continue to the second stage where 42 patients will be assessed for safety and efficacy as part of a phase II study (including the first 14 patients in the phase I study).

Efficacy will be assessed based on local disease control in the lungs and liver, time to systemic disease progression, and overall survival. Patients will be followed for at least 6 months after the last course of NovoTTF-100L is applied to assess survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)
* Stage IV or IIIB with malignant pleural effusion, also locally advanced NSCLC not otherwise amenable to local treatment (surgery or radiotherapy)
* One line of prior chemotherapy
* Measurable disease
* Greater or equal to 18 years
* Life expectancy of at least 12 weeks
* ECOG performance status 0-2
* Laboratory requirements at entry:
* Blood cell counts:
* Absolute neutrophils ≥ 1.0 x 109/L
* Platelets ≥100 x 109/L
* Hemoglobin ≥ 10 g/dl
* Renal function:
* Creatinine clearance ≥ 45 mL/min
* Hepatic functions:
* ASAT and ALAT ≤ 3 x UNL
* Alkaline phosphatase ≤ 5 x UNL
* Signed informed consent prior to start protocol specific requirements
* Pregnancy test (β-HCG) must be negative (needed only for women of childbearing potential).

Exclusion Criteria:

* Known brain metastases or meningeal carcinomatosis
* Other serious concomitant illness of medical conditions:
* Congestive heart failure or angina pectoris except if it is medically controlled.
* Previous history of myocardial infarction within 1 year from study entry.
* Uncontrolled hypertension or arrhythmias
* Implanted pacemaker, defibrillator or deep brain stimulation device
* History of significant neurologic or psychiatric disorders including dementia or seizures
* Active infection requiring iv antibiotics
* Active ulcer, unstable diabetes mellitus or other contra-indication to corticosteroid therapy
* Concurrent treatment with other experimental drugs
* Participation in clinical trials with other experimental agents within 30 days of study entry
* Psychological, familial, sociological or geographical conditions which don't permit medical follow-up and compliance with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Device related toxicity | until 2 months after treatment termination

SECONDARY OUTCOMES:
Time to progression | Six months after recruitment of the last patient in the trial

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Pless, MD, Principal Investigator — Kantonspital Winterthur
Locations (4):
- Switzerland (4):
  - CCRC, Basel
  - Kantonspital Graubunden, Chur
  - Kantonspital Fribourg, Fribourg
  - Kantonspital Winterthur, Winterthur

REFERENCES:
- [Background] Kirson ED, Gurvich Z, Schneiderman R, Dekel E, Itzhaki A, Wasserman Y, Schatzberger R, Palti Y. Disruption of cancer cell replication by alternating electric fields. Cancer Res. 2004 May 1;64(9):3288-95. doi: 10.1158/0008-5472.can-04-0083. PMID 15126372
- [Background] Kirson ED, Dbaly V, Tovarys F, Vymazal J, Soustiel JF, Itzhaki A, Mordechovich D, Steinberg-Shapira S, Gurvich Z, Schneiderman R, Wasserman Y, Salzberg M, Ryffel B, Goldsher D, Dekel E, Palti Y. Alternating electric fields arrest cell proliferation in animal tumor models and human brain tumors. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):10152-7. doi: 10.1073/pnas.0702916104. Epub 2007 Jun 5. PMID 17551011
- [Background] Salzberg M, Kirson E, Palti Y, Rochlitz C. A pilot study with very low-intensity, intermediate-frequency electric fields in patients with locally advanced and/or metastatic solid tumors. Onkologie. 2008 Jul;31(7):362-5. doi: 10.1159/000137713. Epub 2008 Jun 24. PMID 18596382